CLINICAL TRIAL: NCT05432843
Title: A Randomized Controlled Trial Comparing Pregabalin and Placebo in Patients With Persistent Globus Sensation
Brief Title: Comparing Pregabalin and Placebo in Patients With Persistent Globus Sensation
Acronym: Lyrica
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, PI, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S52107
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Globus Sensation
MeSH Terms: conditions — Globus Sensation | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Parallel design with open label period
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the parallel period, the trial is double blinded. After this blinded treatment period, the code will be broken so that patients which received placebo are able to receive the treatment for another 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin (Active Comparator): Treatment with pregabalin in the treatment of globus sensation
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Treatment with placebo in the treatment of globus sensation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Patients receive for one week Pregabalin 75 mg and 7 weeks Pregabalin 150 mg
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — Patients receive a treatment with placebo for 8 weeks
  Arms: Placebo

SUMMARY:
To evaluate the relative merits, safety and effectiveness of pregabalin in globus patients compared with placebo.

DETAILED DESCRIPTION:
Globus, defined as a feeling of a lump in the throat, unexplained by structural lesions, GERD, or histopathology-based esophageal motility disorders, is a frequently occurring symptom of unknown etiology. Today there is no appropriate treatment for patients with a globus sensation. Pathophysiological mechanisms that have been implicated in the pathogenesis of globus include gastroesophageal reflux disease, oesophageal motor disorders, overactive cricopharyngeal muscle, psychological factors, gastric islet patches in the proximal esophagus and deformations of the cervical spine. However, none of these convincingly explains the clinical picture in globus patients.

Investigators recently observed that a large majority (80%) of patients with persistent globus sensation have a pathological EMG examination of the larynx, indicative of neuropathy in the laryngeal area. The investigators believe that this neuropathy may explain some of the symptoms that are experienced by patients with globus, and may actually contribute to some observations of unclear pathophysiological relevance such as a hyperreactive ciricopharyngeal muscle. Neuropathies may respond to specific therapies, such as the pregabalin.

The aim of the study is to evaluate if treatment with pregabalin (Lyrica®) is effective in these patients. The effect of gabapentin, another anti-epileptic drug with therapeutic efficacy in neuropathy, was evaluated in patients with chronic cough as sign of laryngeal sensory neuropathy. In this study 68% of the patients experienced improvement, with an even higher efficacy in the group of patients with a pathological EMG (80%).

In order to better understand the underlying pathophysiology, and how this responds to therapy, the investigators will also evaluate upper esophageal sphincter high resolution manometric properties during the study. An elevated resting pressure in the upper sphincter was already reported in previous studie, but not confirmed in a more recent study, which did report a hyperreactive UES, mainly characterized by a hyperdynamic respiratory pressure change.

Esophageal inlet patches have also been implicated in the pathogenesis of globus, although the exact mechanism remains unclear. In the present study, all patients will undergo a strict evaluation of the upper part of the esophagus during endoscopy, to document presence or absence of inlet patches.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Globus symptoms for more than three months
* First symptoms > 6 months ago
* Signed informed consent

Exclusion Criteria:

* Gabapentin/pregabalin treatment
* Unstable neuroleptic or antidepressive treatment (stable dose during min 8 weeks)
* Symptom relief under PPI treatment (min 8 weeks full dose)
* Patients with persisting esophagitis of Los Angeles grade B or higher under PPI on upper GI endoscopy
* Primary esophageal motility disorder (achalasia, scleroderma, dermatomyositis, …)
* Eosinophilic esophagitis
* Candida esophagitis
* Mechanical explanation of symptoms (e.g. stricture in the pharyngo-esophageal region)
* Pregnancy or plans for pregnancy in the next 12 months (in females)
* History of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-03-12 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 8 weeks
  Proportion of patients in clinical remission or improvement after 8 weeks defined by the Glasgow Edinburgh Throat Scale question 12 ("At present, how annoying do you find your throat sensation?") Ranging from 0-7, where 7 is a worse outcome. Clinical remission is defined as scoring a 0 or 1 on this question.

SECONDARY OUTCOMES:
GETS overall scores | 8 weeks
  Improvement of Glasgow Edinburgh Throat Scale (GETS) overall scores compared between both groups will be evaluated after 8 weeks. The total GETS score is 70, the higher the score, much worse are the symptoms.
Clinical remission | 4 weeks
  Proportion of patients in clinical remission or improvement after 4 weeks defined by the Glasgow Edinburgh Throat Scale question 12 ("At present, how annoying do you find your throat sensation?") Ranging from 0-7, where 7 is a worse outcome. Clinical remission is defined as scoring a 0 or 1 on this question.
GETS overall scores | 4 weeks
  Improvement of Glasgow Edinburgh Throat Scale overall scores compared between both groups will be evaluated after 4 weeks. The total GETS score is 70, the higher the score, much worse are the symptoms.
Overall Treatment Efficacy | 8 weeks
  The Overall Treatment Efficacy evaluation will be analysed by considering the score at 8 weeks. Ranging from 0-6, where 6 is a lower treatment efficacy.
Weekly GETS overall scores | week 1, week 2, week 3, week 4, week 5, week 6, week 7 and week 8
  Improvement of Glasgow Edinburgh Throat Scale overall scores compared between both groups evaluated for each week during the treatment period. Ranging from 0-7, where 7 is a worse outcome. Clinical remission is defined as scoring a 0 or 1 on this question.

OTHER OUTCOMES:
Correlations | 8 weeks
  The correlation between Hospital Anxiety Depression Scale scores, Patient Health Questionnaires scores and therapeutic response evaluated at 8 weeks.
Correlation questionnaires and neuropathy | 8 weeks
  The correlation between Hospital Anxiety Depression Scale scores, Patient Health Questionnaires scores and neuropathy will be evaluated at 8 weeks. The higher score on the Hospital Anxiety Depression Scale and Patient Health Questionnaire, the worse the patients are feeling: more depressed and more anxious and more somatic complaints.
The impact on upper esophageal manometry. | 8 weeks
  The impact of active or placebo treatment on manometry at 8 weeks. Specific upper esophageal manometry parameters are not yet defined.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University Hospital Leuven, Leuven, België
  - Annelies Geeraerts, Leuven

IPD SHARING:
Plan to Share IPD: Undecided